CLINICAL TRIAL: NCT02239926
Title: Effect of Ranolazine on Gastrointestinal Motor Function and Pain in Patients With Diarrhea-predominant Irritable Bowel Syndrome (IBS-D)
Brief Title: Effect of Ranolazine on Gastrointestinal Motor Function and Pain in Patients With IBS-D
Acronym: Ranolazine
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Difficulty in enrolling subjects
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Yuri A. Saito Loftus, Associate Professor of Medicine, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 14-000581
Record Dates: First submitted 2014-09-11; First posted 2014-09-15 (Estimated); Results first posted 2016-02-08 (Estimated); Last update posted 2016-03-15 (Estimated); Status verified 2016-02

CONDITIONS: Diarrhea Predominant Irritable Bowel Syndrome
Keywords: IBS-D
MeSH Terms: interventions — Ranolazine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ranolazine (Active Comparator): tablet, 1000 mg twice daily for four weeks
  Interventions: Drug: Ranolazine
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ranolazine — On January 31, 2006, ranolazine was approved for use in the United States by the Food and Drug Administration (FDA) for the treatment of chronic angina pectoris.
  Other Names: Trade name Ranexa by Gilead Sciences.
  Arms: Ranolazine
Drug: Placebo
  Arms: Placebo

SUMMARY:
Will Ranolazine improve bowel function and abdominal pain in human subjects with IBS-D?

DETAILED DESCRIPTION:
This is a randomized double-blind placebo-controlled pilot study that will use validated bowel questionnaires to evaluate the effects of ranolazine administered orally twice daily in patients with diarrhea predominant IBS (IBS-D). The study will consist of a 2 week run in period, followed by 4 weeks of treatment period with oral ranolazine 1000 mg twice daily. Primary endpoint of the study will be the average Bowel Symptom Scale (BSS) scores for diarrhea and adequate relief of IBS pain and discomfort are secondary end points.

ELIGIBILITY:
Inclusion Criteria

* Males and non-pregnant, non-breastfeeding females with established diagnosis of IBS-D by modified Rome III criteria (Abdominal Pain Intensity: weekly average of worst daily score of >3.0 on a 0 to 10 point scale and Stool Consistency: at least one stool with a consistency of Type 5, 6 or 7 Bristol stool score on at least 2 days per week)
* 18-70 years old
* U.S. resident
* English-speaking (to provide consent and complete questionnaires)

Exclusion Criteria

* Structural or metabolic diseases/conditions that affect the gastrointestinal system
* Unable to withdraw the following medications 48 hours prior to the study:

  * Drugs that alter GI transit including Lomotil, and bile acid binders such as cholestyramine, prokinetics (e.g. metoclopramide, cisapride and erythromycin), narcotics (e.g. oxycodone, morphine) and anticholinergics (dicyclomine, hyoscyamine).
  * Analgesic drugs including narcotics, NSAID, cyclooxygenase-2 ( COX2) inhibitors (celecoxib, rofecoxib, and valdecoxib)
  * GABAergic agents (baclofen)
  * Benzodiazepines (e.g. lorazepam, alprazolam, and diazepam). Low stable doses of thyroid replacement, estrogen replacement, and low dose aspirin for cardioprotection and birth control pills or depot injections are permissible.
* Unable to withdraw the following medications, which are contraindications of ranolazine:

  * Strong Cytochrome P450, Family 3, Subfamily A (CYP3A) inhibitors (e.g. ketoconazole, clarithromycin, and nelfinavir)
  * CYP3A inducers (e.g. rifampin, phenobarbital, St. John's wort)
* Female subjects who are pregnant or breastfeeding.
* Current symptoms of severe depression, as measured by Hospital Anxiety And Depression Scale ( HADS) score greater than 15.
* Clinical evidence (including physical exam, ECG, laboratory studies and review of the medical history) of significant cardiovascular, respiratory, renal, hepatic, gastrointestinal, hematological, neurological, psychiatric, or other disease that interfere with the objectives of the study.
* The Corrected QT Interval (QTc) > 490 msec.
* Active alcoholics not in remission or known substance abusers.
* Liver cirrhosis
* Patients with clinically significant hepatic disease.
* Major cardiovascular events in the last 6 months.
* Participation in another clinical trial (within 30 days).
* Incarcerated.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2014-09; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yuri A Saito, MD,MPH, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled at Mayo Clinic, Rochester Minnesota.
Pre-assignment Details: 2 subjects were screen failures and were not randomized.
  1 subject signed informed consent, but the study was suspended prior to that subject's randomization.
Period: Overall Study
Arm/Group | Ranolazine | Placebo
Started | 0 | 2
Completed | 0 | 1
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ranolazine | Placebo | Total
Number analyzed (Participants) | 0 | 2 | 2
Age, Categorical [Number; unit: participants]
  <=18 years |  | 0 | 0
  Between 18 and 65 years |  | 2 | 2
  >=65 years |  | 0 | 0
Gender [Number; unit: participants]
  Female |  | 2 | 2
  Male |  | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States |  | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Diarrhea Using the Bowel Symptom Score (BSS).
Description: BSS is a 100-mm visual analog scale for each symptom of Irritable Bowel Syndrome (IBS) (pain or discomfort, bloating, and diarrhea) with an overall severity score. Lower scores indicate symptoms are not present and higher scores indicate severe symptoms.
Time Frame: baseline to 4 weeks
Population: The one subject who completed the study did not have complete data, so no analysis was performed. Study was terminated due to difficulty with enrollment.
Arm/Group | Ranolazine | Placebo
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Mean Abdominal Pain
Description: Daily abdominal pain intensity was rated using an 11-point (0-10) numeric rating scale, with 0 being no pain, and 10 being the worst pain imaginable. Participants were asked to rate their worst abdominal pain over the past 24 hours.
Time Frame: baseline to 4 weeks
Population: as for outcome 1
Arm/Group | Ranolazine | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Ranolazine | Placebo
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/2
Other Adverse Events (participants affected / at risk) | 0/0 | 0/2

LIMITATIONS AND CAVEATS:
The study was terminated early due to enrollment issues.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes